CLINICAL TRIAL: NCT03263091
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Investigating the Efficacy and Safety of Roxadustat (FG-4592) for Treatment of Anemia in Patients With Lower Risk Myelodysplastic Syndrome (MDS) With Low Red Blood Cell (RBC) Transfusion Burden (LTB)
Brief Title: Efficacy and Safety of Roxadustat for Treatment of Anemia in Participants With Lower Risk Myelodysplastic Syndrome With Low Red Blood Cell Transfusion Burden
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study did not meet its primary efficacy endpoint.
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-4592-082
Record Dates: First submitted 2017-08-22; First posted 2017-08-28 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Primary MDS (Very Low, Low or Intermediate IPSS-R With <5% Blasts); Anemia
Keywords: Myelodysplastic Syndromes; Anemia; Hemoglobin (Hb); Low Risk Myelodysplastic Syndrome; Low Risk MDS
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Open-label, lead-in: Participants will receive sequential escalating roxadustat doses (1.5 milligrams/kilograms [mg/kg], 2.0 mg/kg and 2.5 mg/kg), three times a week (TIW) based upon their actual weight at the randomization visit to identify the starting dose for double-blind period.
  Double-blind: Participants will receive roxadustat 2.5 mg/kg TIW based upon their body weight for a duration of 52 weeks.
  Open-label: Participants with high serum erythropoietin levels (>400 milli-international units [mIU]/milliliter [mL] mIU/mL) will receive roxadustat 2.5 mg/kg TIW based upon their body weight for a duration of 52 weeks.
  Interventions: Drug: Roxadustat
- Placebo (Placebo Comparator): Double-blind: Participants will receive placebo matching to roxadustat for a duration of 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roxadustat — Oral tablets
  Other Names: FG-4592; ASP1517; AZD9941
  Arms: Roxadustat
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether FG-4592 is safe and effective in the treatment of anemia in participants with lower risk MDS and low red blood cell transfusion burden.

DETAILED DESCRIPTION:
This study includes an Open-Label Lead in, a Double-Blind component, and an Open-Label High Erythropoietin component. There is a screening period of up to 42 days followed by a treatment period of 52 weeks and a 4-week end of treatment assessment.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of primary MDS classified by the International Prognostic Scoring System - Revised (IPSS-R) as very low, low or intermediate risk with <5% bone marrow blasts. There is no minimum time from diagnosis to registration/randomization except to allow for proper IPSS-R classification to be made (within 16 weeks prior to randomization), and to show transfusion dependence for participants in both portions of the study.
* RBC transfusion of either 2-4 pRBC units during the 8 weeks prior to registration/randomization or 1 pRBC in two consecutive periods of 8 weeks within the 16 weeks prior to registration/randomization. Open-Label Lead-in participants only, the requirement to demonstrate transfusion dependence can also be met by a Principal Investigator starting this particular participant on pRBC transfusion during the screening period.
* No restriction on prior use of recombinant erythropoietins or analogues (erythropoiesis-stimulating agents [ESAs]), except no ESA use within 8 weeks prior to Day 1 registration/randomization.
* Hemoglobin (Hb) ≤10.0 grams/deciliter (g/dL) during screening
* Eastern Cooperative Oncology Group (ECOG) of 0-2 at screening

Key Exclusion Criteria:

* Diagnosis of secondary MDS associated with prior chemotherapy, extensive radiation therapy (>25% of bone marrow reserve), and or/other significant chemical or radiation exposure
* Significant myelofibrosis (>2+ fibrosis)
* MDS associated with 5q(del) cytogenetic abnormality
* Screen serum erythropoietin level > 400 milli-international units (mIU)/milliliter (mL) • Clinically significant anemia, as determined by the investigator, due to non-MDS etiologies such as iron deficiency, vitamin B12 or folate deficiency, autoimmune or hereditary hemolysis or anemia or hemorrhage or hereditary anemia such as sickle cell anemia or thalassemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (111):
- United States (28):
  - Investigational Site, Bakersfield, California
  - Investigational Site, Beverly Hills, California
  - Investigational Site, Burbank, California
  - Investigational Site, Encino, California
  - Investigational Site, Laguna Hills, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Oceanside, California
  - Investigational Site, Pasadena, California
  - Investigational Site, Santa Maria, California
  - Investigational Site, Torrance, California
  - Investigational Site, Valencia, California
  - Investigational Site, Ventura, California
  - Investigational Site, Westlake Village, California
  - Investigational Site, Whittier, California
  - Investigational Site, Grand Junction, Colorado
  - Investigational Site, Pembroke Pines, Florida
  - Investiational Site, Weston, Florida
  - Investgational site, Atlanta, Georgia
  - Investigational Site, Augusta, Georgia
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Canton, Ohio
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Mayfield Heights, Ohio
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Charleston, South Carolina
  - Investigational Site, Houston, Texas
  - Investigational Site, Charlottesville, Virginia
- Australia (5):
  - Investigational Site, Darlinghurst, New South Wales
  - Investigational Site, Liverpool, New South Wales
  - Investigational Site, South Brisbane, Queensland
  - Investigational Site, Victoria Park, Saint Albans
  - Investigational Site, Hobart, Tasmania
- Belgium (6):
  - Investigational Site, Wilrijk, Antwerpen
  - Investigational Site, Brussels, Brussels Capital
  - Investigational Site, Hasselt, Limburg
  - Investigational Site, Bruges, West-Vlaanderen
  - Investigational Site, Brussels
  - Investigational Site, Yvoir
- Canada (2):
  - Investigational Site, Vancouver, British Columbia
  - Investigational Site, London, Ontario
- Investigational Site, Odense, Denmark
- France (4):
  - Investigational Site, Nice, Alpes-Maritimes
  - Investigational Site, Grenoble, Isère
  - Investigational Site, Paris
  - Investigational Site, Tours
- Germany (6):
  - Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Investigational Site, München, Bavaria
  - Investigational Site, Münster, North Rhine-Westphalia
  - Investigational Site, Dresden, Saxony
  - Investigational Site, Leipzig, Saxony
  - Investigational Site, Düsseldorf
- India (2):
  - Investigational Site, Vellore, Tamil Nadu
  - Investigational Site, Kolkata, West Bengal
- Israel (7):
  - Investigational Site, Kfar Saba, Central District
  - Investigational Site, Ẕerifin, Central District
  - Investigational Site, Nahariya, Northern District
  - Investigational Site, Haifa
  - Investigational Site, Ramat Gan
  - Investigational Site, Tel Aviv
  - Investigational site, Tel Litwinsky
- Italy (14):
  - Investigational Site, Monza, Lombardy
  - Investigational Site, Meldola, Ravenna
  - Investigational Site, Alessandria
  - Investigational Site, Bologna
  - Investigational Site, Florence
  - Investigational Site, Genova
  - Investigational Site, Lecce
  - Investigational Site, Milan
  - Investigational Site, Reggio Calabria
  - Investigational Site, Rimini
  - Investigational Site, Roma
  - Investigational Site, Terni
  - Investigational Site, Torino
  - Investigational Site, Varese
- Poland (7):
  - Investigational Site, Bialystok
  - Investigational Site, Bydgoszcz
  - Investigational Site, Krakow
  - Investigational Site, Piła
  - Investigational Site, Skorzewo
  - Investigational Site, Słupsk
  - Investigational Site, Warsaw
- Russia (5):
  - Investigational Site, Kaluga, Russian Federation
  - Investigational Site, Moscow, Russian Federation
  - Investigational Site, Omsk, Russian Federation
  - Investigational Site, Saint Petersburg, Russian Federation
  - Investigational Site, Saint Petersburg
- South Korea (5):
  - Investigational Site, Incheon, Incheon Gwang'yeogsi
  - Investigational Site, Incheon, Incheon Gwangyeogsi
  - Investigational Site, Hwasun, Jeonranamdo
  - Investigational Site, Seoul, Seoul Teugbyeolsi
  - Investigational Site, Seoul
- Spain (8):
  - Investigational Site, Sabadell, Barcelona
  - Investigational Site, Barcelona, Catalonia
  - Investigational Site, Pamplona, Navarre
  - Investigational Site, Barcelona
  - Investigational Site, Madrid
  - Investigational Site, Salamanca
  - Investigational Site, Seville
  - Investigational Site, Valencia
- Turkey (Türkiye) (6):
  - Investigational Site, Ankara
  - Investigational Site, Dikimevi
  - Investigational Site, Izmir
  - Investigational Site, Kayseri
  - Investigational Site, Tekirdağ
  - Investigational Site, Yenişehir
- United Kingdom (5):
  - Investigational Site, Boston, Lincolnshire
  - Investigational Site, Headington, Oxford
  - Investigational Site, Harrow
  - Investigational Site, London
  - Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henry DH, Glaspy J, Harrup R, Mittelman M, Zhou A, Carraway HE, Bradley C, Saha G, Modelska K, Bartels P, Leong R, Yu KP. Roxadustat for the treatment of anemia in patients with lower-risk myelodysplastic syndrome: Open-label, dose-selection, lead-in stage of a phase 3 study. Am J Hematol. 2022 Feb 1;97(2):174-184. doi: 10.1002/ajh.26397. Epub 2021 Nov 9. PMID 34724251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 3 components: Open-label (OL) Lead-in, Double-blind (DB), and OL High-erythropoietin (High-EPO) component.
Pre-assignment Details: Participants were enrolled in sequential dose level cohorts in OL lead-in component prior to the start of DB component. Concurrent with enrollment in DB component, participants with high serum EPO levels (>400 milli-international units [mIU]/milliliter [mL]), exclusionary for DB component, were enrolled in an OL high-EPO component. Participants with lower-risk myelodysplastic syndrome (MDS) with low transfusion burden (LTB) were randomized 3:2 to roxadustat or matching placebo in DB component.
Groups:
- OL Component (Cohort 1): Roxadustat 1.5 mg/kg: Participants received roxadustat 1.5 milligrams (mg)/kilograms (kg), three times a week (TIW) for 52 weeks.
- OL Component (Cohort 2): Roxadustat 2.0 mg/kg: Participants received roxadustat 2.0 mg/kg, TIW for 52 weeks.
- OL Component (Cohort 3): Roxadustat 2.5 mg/kg: Participants received roxadustat 2.5 mg/kg, TIW for 52 weeks.
- OL High-EPO Component: Roxadustat 2.5 mg/kg: Participants with high serum EPO levels (>400 mIU/mL) received roxadustat 2.5 mg/kg TIW for 52 weeks.
- DB Component: Roxadustat: Participants received roxadustat 2.5 mg/kg TIW for 52 weeks.
- DB Component: Placebo: Participants received placebo matched to roxadustat for 52 weeks.
Period: OL Component
Arm/Group | OL Component (Cohort 1): Roxadustat 1.5 mg/kg | OL Component (Cohort 2): Roxadustat 2.0 mg/kg | OL Component (Cohort 3): Roxadustat 2.5 mg/kg | OL High-EPO Component: Roxadustat 2.5 mg/kg | DB Component: Roxadustat | DB Component: Placebo
Started | 8 | 8 | 8 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 8 | 8 | 8 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 0 | 0 | 0
Not Completed | 2 | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Period: OL High-EPO Component
Arm/Group | OL Component (Cohort 1): Roxadustat 1.5 mg/kg | OL Component (Cohort 2): Roxadustat 2.0 mg/kg | OL Component (Cohort 3): Roxadustat 2.5 mg/kg | OL High-EPO Component: Roxadustat 2.5 mg/kg | DB Component: Roxadustat | DB Component: Placebo
Started | 0 | 0 | 0 | 20 | 0 | 0
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 20 | 0 | 0
Completed | 0 | 0 | 0 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 10 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 3 | 0 | 0
Period: DB Component
Arm/Group | OL Component (Cohort 1): Roxadustat 1.5 mg/kg | OL Component (Cohort 2): Roxadustat 2.0 mg/kg | OL Component (Cohort 3): Roxadustat 2.5 mg/kg | OL High-EPO Component: Roxadustat 2.5 mg/kg | DB Component: Roxadustat | DB Component: Placebo
Started | 0 | 0 | 0 | 0 | 82 | 58
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 82 | 58
Completed | 0 | 0 | 0 | 0 | 38 | 37
Not Completed | 0 | 0 | 0 | 0 | 44 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 22 | 8
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 7 | 4
Not completed — Other than specified | 0 | 0 | 0 | 0 | 8 | 6

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- OL Component (Cohort 1): Roxadustat 1.5 mg/kg: Participants received roxadustat 1.5 mg/kg, TIW for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | OL Component (Cohort 1): Roxadustat 1.5 mg/kg | OL Component (Cohort 2): Roxadustat 2.0 mg/kg | OL Component (Cohort 3): Roxadustat 2.5 mg/kg | OL High-EPO Component: Roxadustat 2.5 mg/kg | DB Component: Roxadustat | DB Component: Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 20 | 82 | 58 | 184
Age, Customized [Count of Participants; unit: Participants]
  <65 Years | 3 | 0 | 2 | 8 | 18 | 14 | 45
  ≥65 Years | 5 | 8 | 6 | 12 | 64 | 44 | 139
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 6 | 36 | 21 | 75
  Male | 5 | 5 | 2 | 14 | 46 | 37 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 1 | 2 | 6
  Not Hispanic or Latino | 7 | 7 | 6 | 19 | 78 | 55 | 172
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 3 | 14 | 7 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 8 | 8 | 17 | 63 | 49 | 152
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 5 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: OL and OL High-EPO Components: Number of Participants Who Achieved Red Blood Cell (RBC) Transfusion Independence (TI) ≥8 Weeks (≥56 Consecutive Days) Since First Dose in the First 28 Weeks of Treatment
Description: The RBC TI was defined as the absence of any intravenous (IV) RBC transfusion (packed cell or whole blood) during any consecutive 56 days during the treatment period. Data presented is for number of participants with RBC TI ≥8 weeks (≥56 consecutive days) since first dose in the first 28 weeks of treatment.
Time Frame: 28 weeks
Population: The full analysis set (FAS) included all enrolled participants who received at least 1 dose of study medication, and at least 1 corresponding on-treatment hemoglobin (Hb) assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | OL Component (Cohort 1): Roxadustat 1.5 mg/kg | OL Component (Cohort 2): Roxadustat 2.0 mg/kg | OL Component (Cohort 3): Roxadustat 2.5 mg/kg | OL High-EPO Component: Roxadustat 2.5 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 20
Participants | 3 | 1 | 5 | 3

2. Primary Outcome: DB Component: Number of Participants Who Achieved RBC TI ≥56 Consecutive Days Since First Dose in the First 28 Weeks of Treatment
Description: RBC TI was defined as the absence of any IV RBC transfusion (packed cell or whole blood) during any consecutive 56 days during the treatment period. Data presented is for number of participants with RBC TI ≥56 consecutive days since first dose in the first 28 weeks of treatment.
Time Frame: 28 weeks
Population: FAS included all enrolled participants who received at least 1 dose of study medication, and at least 1 corresponding on-treatment Hb assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 80 | 57
Participants | 38 | 19
Statistical Analysis 1: Comparison: DB Component: Roxadustat vs DB Component: Placebo; The odds ratio along with its 95% confidence interval (CI) were calculated based on the Cochran-Mantel-Haenszel (CMH) chi-square test adjusting for the stratification factors (EPO level, International Prognostic Scoring System - Revised [IPSS-R] risk category and RBC transfusion burden); Test type: Other; p = 0.217, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.582, 95% CI 2-sided [0.761 to 3.290]

3. Secondary Outcome: OL and OL High-EPO Components: Number of Participants Who Achieved TI ≥50% Reduction From Baseline in Number of Packs of Red Blood Cells (pRBC) Transfusions Over 8 Weeks
Description: Number of pRBC transfusions at baseline was defined as pRBC transfusions requirement during 8-week period prior to the start of first study medication. Responders were defined as participants with at least a 50% reduction in the number of pRBC transfusions over any 8-week (56 consecutive days) period during the study as compared with the baseline.
Time Frame: Baseline up to Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | OL Component (Cohort 1): Roxadustat 1.5 mg/kg | OL Component (Cohort 2): Roxadustat 2.0 mg/kg | OL Component (Cohort 3): Roxadustat 2.5 mg/kg | OL High-EPO Component: Roxadustat 2.5 mg/kg
Number analyzed (Participants) | 8 | 8 | 8 | 20
Participants | 5 | 3 | 7 | 8

4. Secondary Outcome: DB Component: Number of Participants Who Achieved TI ≥56 Consecutive Days Since First Dose in 52 Weeks of Treatment
Description: RBC TI was defined as the absence of any IV RBC transfusion (packed cell or whole blood) during any consecutive 56 days during the treatment period. Data presented is for number of participants with RBC TI ≥56 consecutive days since first dose in the 52 weeks of treatment.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 80 | 57
Participants | 44 | 23

5. Secondary Outcome: DB Component: Number of Participants Who Achieved TI ≥56 Consecutive Days Anytime During the Study
Description: RBC TI was defined as the absence of any IV RBC transfusion (packed cell or whole blood) during any consecutive 56 days anytime during the study (up to Week 56).
Time Frame: Baseline up to Week 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 80 | 57
Participants | 52 | 29

6. Secondary Outcome: DB Component: Number of Participants Who Achieved ≥50% Reduction From Baseline in Number of pRBC Transfusions Over 8 Weeks
Description: Baseline number of transfusions (pRBC/8-weeks) = total number of packs of rRBCs within 16 weeks prior to first dose/2. A pRBC transfusion reduction responder was defined as a participant who achieved ≥50% reduction in number of pRBC transfusions over 8 weeks compared to their baseline for any 8 week period in the duration begining with the first dose date (Day 1) and ending with the end of study or treatment discontinuation due to adverse event (AE)/serious adverse event (SAE) or death, whichever came earlier.
Time Frame: Baseline up to Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 80 | 57
Participants | 59 | 37

7. Secondary Outcome: DB Component: Cumulative Number of Participant Exposure Weeks (PEW) of TI Over the First 28 Weeks of Treatment
Description: The PEW of TI periods over the first 28 weeks was added up to a cumulative number of weeks. For a participant with at least 1 TI response period over the first 28 weeks, the last TI response period was ended with the date of a subsequent RBC transfusion, visit date at Week 28, date of the end of study or treatment discontinuation due to AE/SAE or death, whichever came earlier. For a participant with no TI response period over the first 28 weeks, the cumulative number of PEW was set to zero.
Time Frame: 28 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 80 | 57
weeks | 9.60 (11.537) | 7.60 (11.557)

8. Secondary Outcome: DB Component: Change From Baseline in Number of pRBC Packs Transfused Over the First 28 Weeks of Treatment
Description: Number of pRBC transfusions at baseline was defined as pRBC transfusions requirement during 8-week period prior to the start of first study medication.
Time Frame: Baseline, Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pRBC packs
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 80 | 57
pRBC packs | -0.13 (2.314) | 0.44 (1.833)

9. Secondary Outcome: DB Component: Number of Participants Who Achieved TI ≥20 Consecutive Weeks During the Study
Description: ≥20 consecutive weeks TI was defined as the absence of any IV RBC transfusion (packed cell or whole blood) during any consecutive 140 days anytime during the study (up to 56 weeks). TI was estimated between the first dose date (Day 1) and the end of study (Week 56) or treatment discontinuation due to AE/SAE or death, whichever came earlier.
Time Frame: Baseline up to Week 56
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 80 | 57
Participants | 23 | 15

10. Secondary Outcome: DB Component: Mean Change From Baseline in the Patient-Reported Outcomes Measurement Information System-Short Form (PROMIS-SF) v2.0 Physical Function (PF) 10b Score at Week 9
Description: The PROMIS physical function item measures self-reported, current capability to carry out activities that require physical actions, ranging from self-care (activities of daily living) to more complex activities that require a combination of skills, often within a social context. The PF 10-item short form which contains 10 questions was used in this study, and each item was scored on a 5-point rating scale (1 [unable to do] to 5 [without any difficulty]), with higher scores indicating better functioning. Total raw score was the sum of the response to each question, with the lowest possible raw score 10 (poor physical function) and the highest possible raw score 50 (better physical function). Raw scores converted to T-scores (as detailed in the T-score conversion table for PROMIS-SF v2.0 Physical Function 10b) with a mean of 50 and a standard deviation (SD) of 10. T-scores ranged from minimum 13.8 to maximum 61.3 possible scores with higher scores indicating better physical functioning.
Time Frame: Baseline, Week 9
Population: FAS included all enrolled participants who received at least 1 dose of study medication, and at least 1 corresponding on-treatment Hb assessment. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 71 | 52
T-score | -1.9 (7.29) | -0.4 (6.77)

11. Secondary Outcome: DB Component: Mean Change From Baseline in the PROMIS-SF v1.0 Fatigue 13a Score at Week 9
Description: Fatigue was measured using the 13-item fatigue scale of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System, each item was scored on a 5-point rating scale ranging from 1 "not at all" to 5 "very much", with lower scores indicating better functioning. Total raw score was the sum of the response to each question, with the lowest possible raw score 13 (lowest level of fatigue) and the highest possible raw score 65 (highest level of fatigue), with lower scores indicating better functioning. Raw scores converted to T-scores (as detailed in the T-score conversion table for PROMIS-SF v1.0 Fatigue 13a) with a mean of 50 and a SD of 10. T-scores ranged from minimum 30.3 to maximum 83.5 possible scores with lower scores indicating better functioning.
Time Frame: Baseline, Week 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 67 | 52
T-score | 1.9 (7.61) | -0.6 (7.36)

12. Secondary Outcome: DB Component: Mean Change From Baseline in the European Quality of Life Five Dimensional Five Level Health Questionnaire (EQ-5D-5L) Visual Analogue Scale Score at Week 9
Description: The EQ-5D questionnaire is designed for self-completion by participants. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problem, moderate problems, severe problems, and unable to/extreme problems. The questionnaire also included a visual analogue scale, where the participant was asked to rate current health status on a scale of 0-100, with 0 being the worst imaginable health state and 100 being the best imaginable health.
Time Frame: Baseline, Week 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Component: Roxadustat | DB Component: Placebo
Number analyzed (Participants) | 71 | 55
units on a scale | -1.7 (20.31) | 1.6 (16.18)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 56
Description: The safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | OL Component (Cohort 1): Roxadustat 1.5 mg/kg | OL Component (Cohort 2): Roxadustat 2.0 mg/kg | OL Component (Cohort 3): Roxadustat 2.5 mg/kg | OL High-EPO Component: Roxadustat 2.5 mg/kg | DB Component: Roxadustat | DB Component: Placebo
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 3/20 | 7/82 | 4/58
Serious Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 1/8 | 6/20 | 22/82 | 10/58
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8 | 6/8 | 15/20 | 68/82 | 46/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL Component (Cohort 1): Roxadustat 1.5 mg/kg (N=8) | OL Component (Cohort 2): Roxadustat 2.0 mg/kg (N=8) | OL Component (Cohort 3): Roxadustat 2.5 mg/kg (N=8) | OL High-EPO Component: Roxadustat 2.5 mg/kg (N=20) | DB Component: Roxadustat (N=82) | DB Component: Placebo (N=58)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 2 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 4 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 3
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OL Component (Cohort 1): Roxadustat 1.5 mg/kg (N=8) | OL Component (Cohort 2): Roxadustat 2.0 mg/kg (N=8) | OL Component (Cohort 3): Roxadustat 2.5 mg/kg (N=8) | OL High-EPO Component: Roxadustat 2.5 mg/kg (N=20) | DB Component: Roxadustat (N=82) | DB Component: Placebo (N=58)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 5 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 3 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 2 | 0 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 2 | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 6 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 19 | 7
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 6 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 4 | 11 | 7
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 15 | 6
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 2 | 9 | 4
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 5 | 1
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 2 | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 6
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 4 | 5
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 2
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Nasal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 10 | 7
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 3 | 8 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 6 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 2 | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 6 | 5
Folate deficiency (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 4 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 3
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1 | 11 | 10
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 7 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 9 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1 | 8 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 8 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Trichodynia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 4 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study did not meet its primary efficacy endpoint; hence, the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03263091/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03263091/SAP_001.pdf